CLINICAL TRIAL: NCT06316375
Title: Assessment Of STUMBL Score (STUdy of the Management of BLunt Chest Wall Trauma) As A Risk Stratification Tool In Management Of Blunt Chest Trauma Patients In Emergency Departments: A Multicenter Study
Brief Title: STUMBL Score as a Risk Stratification Tool for Management of Blunt Chest Trauma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, hadeer mahmoud saber youssef, Emergency medicine resident, Assiut University
Other Study IDs: STUMBL blunt chest trauma
Record Dates: First submitted 2024-03-03; First posted 2024-03-18 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Blunt Injury of Thorax
Keywords: Blunt chest trauma; STUMBL score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess validity of the STUMBL score in EGYPT for complications of blunt chest trauma without multi-trauma and immediate life-threatening injuries and identify patients at risk of in- hospital mortality or ICU admission and predict survival in both Assiut & Suez Canal University Hospitals.

DETAILED DESCRIPTION:
The STUMBL Score (STUdy of the Management of BLunt chest wall trauma) (also referred to as the Battle score) is a clinical prediction model that was developed and externally validated in 2014 in the UK . The purpose of the model is to assist in the clinical decision-making of patients with blunt chest wall trauma (excluding those with life-threatening injuries) in the Emergency Department (ED), through the calculation of a percentage risk of complications which in turn, provides a recommended discharge disposition. The STUMBL score includes five predictors: age at attendance, number of rib fractures, chronic lung disease, use of pre-injury anticoagulants and oxygen saturation (SpO2). This is the first score to introduce clinical variables, specifically chronic lung disease and anticoagulation, in contrast to other scores which have used anatomical variables and age alone. A huge benefit of the STUMBL score is that these variables are all routinely measured in the ED. Whilst other scores exist, the STUMBL Score is the only externally validated model with excellent predictive capabilities, that can be used for adult patients of all ages with blunt chest trauma presenting to the ED, not just a specific age group or severity of injury.

Collected data will be analyzed and tabulated by using appropriate statistical methods.

Statistical analysis will be performed by the SPSS statistical software computer program version 20 (Statistical Package for Social Science), Medcalc v.11.6.and Open Epi V.3.01.

Data will be described using mean ± standard deviation (SD) and frequencies according if they are quantitative or qualitative respectively.

Parametric tests will be used in the current study if data proved to be normally distributed.

For all statistical tests, a P value less than 0.05 will be taken to indicate a significant difference.

ELIGIBILITY:
Inclusion Criteria:

* The present study will be conducted on patients of blunt chest trauma of both genders "without intently selected certain gender" and had 18 years old or more.

Exclusion Criteria:

* patients <18 years of age
* patients with life threatening conditions

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with blunt chest trauma satisfying inclusion criteria and does not include exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome was to assess the validity of the STUMBL score for all complications of chest blunt trauma, originally defined by the STUMBL authors | 7 days
  These complications include:
  * In-hospital mortality.
  * All pulmonary complications (including but not restricted to haemothorax, pneumothorax, lung contusion, pneumonia, and empyema, excluding rib fractures).
  * Need for ICU admission.
  * Prolonged hospital stay defined as a total hospital stay of 7 days or more

SECONDARY OUTCOMES:
Secondary outcomes validated the STUMBL score using a composite of early and delayed complications. | 72 hours
  Early complications:
  * Presence of a pulmonary complication on arrival to ED as defined above
  * Admission to ICU from ED
  Delayed complications:
  * Delayed pulmonary complications defined as pulmonary complications developing or discovered after discharge from the ED to the ward or community,including lung contusion,pleural effusion,empyema, hemothorax,pneumothorax,pneumomediastinum,pneumonia or pulmonary embolism.
  * Delayed escalation in care,defined as a requirement for ICU admission because of chest trauma related complications at any point after discharge from the ED to the ward or community.
  * Unplanned re-presentation to the ED,Patient discharged from ED on the first presentation but re-presented to ED with complications of chest trauma that was not a planned followup assessment within 72h of discharge for patients whose initial hospital stay was 1day or less (including those discharged directly from ED and those admitted to a ward for less than 2days).